CLINICAL TRIAL: NCT07137455
Title: EDEN Intracardiac Electrogram Recording and Classifying System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10002526; 002526-H
Record Dates: First submitted 2025-08-19; First posted 2025-08-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-08-13

CONDITIONS: Ventricular Arrhythmia
Keywords: intracardiac electrogram; radial depth

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EDEN Intracardiac Electrogram Recording and Classifying System (Experimental): EDEN will be used to record and classify intracardiac electrograms obtained in the practice of medicine.
  Interventions: Device: EDEN Intracardiac Electrogram Recording and Classifying System

INTERVENTIONS:
Device: EDEN Intracardiac Electrogram Recording and Classifying System — EDEN will be used to record and classify intracardiac electrograms obtained in the practice of medicine.

SUMMARY:
Background:

Heart surgeons use electrocardiogram (ECG) machines to record electrical signals from the heart during procedures. Normal ECG machines connect only to the skin. Special ECG machines connect directly to the heart; they are a safer option during procedures. Researchers want to test a new ECG machine called the EDEN system.

Objective:

To test the EDEN system in people having heart procedures. The new system will be used along with an approved special ECG machine.

Eligibility:

People aged 21 years or older who need to have a heart procedure. These procedures can include (1) electrophysiology mapping or ablation; and (2) conduction system pacing.

Design:

Researchers will review participants' medical records. No extra tests are needed.

Participants will have their heart procedure as planned.

The EDEN system will be linked to the special ECG used during the procedure. An extra electrode may be placed on the participant's body. Electrodes are small stickers attached to wires that go to the machine.

The EDEN system will record and analyze electrical signals already being measured. It will not interfere with participants' care. No medical decisions well be made based on its data.

No follow-up visits are needed for this study....

DETAILED DESCRIPTION:
Study Description:

The study tests a hardware electrocardiography appliance used to record and classify intracardiac electrograms obtained in the practice of medicine. No diagnoses or clinical decisions are based on the findings in this study.

Objectives:

The primary objective is to determine whether the classifier accurately identifies the EDEN radial depth category.

Endpoints:

Primary endpoint: The primary endpoint is classifier accuracy.

Exploratory endpoints: Correspondence of EDEN electrograms with CT and CMR findings (of myocardial segmental thickness, scar, and possibly relaxometry); Impact of abnormal conduction, induced or observed during the EP procedure, on EDEN electrogram morphology. Technical success of acquiring and classifying EDEN electrograms.

ELIGIBILITY:
* INCLUSION CRITERIA
* Age >= 21 years
* Undergoing a medically-necessary invasive cardiac electrophysiology mapping and/or ablation procedure for ventricular arrhythmia, or conduction system pacing procedure

EXCLUSION CRITERIA

* Does not consent to participate, or unable to consent to participate
* Hemodynamic instability or emergency procedure

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Classifier accuracy | During intracardiac electrograms procedure
  The primary endpoint is classification accuracy of EDEN electrograms automated classifications compared with operator-determined classifications of radial depth according to a five-element ordinal scale (cameral, subendocardial, midmyocardial, subepicardial, pericardial). Agreement will be assessed using standard metrics such as concordance.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Lederman, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD that underline results in a publication will be shared. Medical images will not be shared because of intrinsic inability to protect confidentiality with reasonable effort.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available by the end of the project or protocol or at the time of associated publication.
Access Criteria: BioData Catalyst is supported by NHLBI and access to data is controlled by the NHLBI Data Access Committee (DAC) utilizing the database of Genotypes and Phenotypes (dbGaP) permissions infrastructure. In order to access controlled-access data in BioData Catalyst, an investigator must have an approved Data Access Request (DAR) in dbGaP.